CLINICAL TRIAL: NCT01439997
Title: Desmopressin Melt Therapy in Nocturnal Polyuria Patients: Pharmacodynamic Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011/567
Record Dates: First submitted 2011-09-14; First posted 2011-09-23 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Nocturia
Keywords: Nocturnal polyuria
MeSH Terms: conditions — Nocturia | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Desmopressin Melt Therapy in Nocturnal Polyuria Patients (Experimental)
  Interventions: Drug: Desmopressin

INTERVENTIONS:
Drug: Desmopressin — Administration of minirin melt 60 µg: desmopressin (acetate) 60 µg oral lyophilisate.
  Other Names: Minirin Melt 60 µg

SUMMARY:
The objective of this study is to find out what the pharmacodynamic (PD) characteristics of desmopressin melt are in nocturia patients (compared to healthy volunteers and children). The main questions the investigators want to answer are:

* Are differences related to the pathophysiological factors involved in nocturia?
* Are there age/gender/size differences?
* Can the investigators identify patients who are likely to develop hyponatraemia?
* Can the investigators individualize treatment and reduce risk for hyponatraemia?

The patient will be given a prescription to buy Minirin Melt 60µg at the local pharmacy. During 30 days, the patient has to take Minirin Melt 60µg in the evening before going to bed.

There are two groups of patients:

Group A:

Patients that still have to undergo an evaluation phase, according to standard procedures (e.g. osmolality test, blood sample). This procedure is not a part of this study. The study starts when the 1st Minirin Melt tablet has been taken (= day 1).

Group B:

This group already went through the evaluation phase (by participation to study 1 or study 3 as mentioned above) and they have been prescribed Minirin Melt 60 µg ambulatory.

The study starts when the patients takes his first prescribed Minirin Melt tablet:

* On day 3 and day 7 a blood sample will be taken at the UZ Ghent for safety control (Na+, K+, creatinin, osmolality = good clinical practice guideline). These first 2 visits (day 3 and day 7) are standard procedure. If the patient is at high risk for side effects, blood has to be taken during the first 7 days.
* On day 3 the patient has to give a urine sample.
* Patients have to fill out a frequency/volume chart during the first 14 days.
* On day 30, a 3rd blood sample will be taken

ELIGIBILITY:
Inclusion Criteria:

* written informed consent prior to the performance of any study-related activity
* patients, men and women, 18 years and older, with an average of ≥ 2 nocturnal voids per night
* evidence for nocturnal polyuria (nocturnal urine volume >33% of total volume over 24h), determined on frequency/volume chart
* Diuresis <2.5L

Exclusion Criteria:

* hypersensitivity/anaphylactic reaction on desmopressin or one of the other substances
* pregnancy
* genitourinary tract pathology (infection, tumor,...)
* urolithiasis
* suspicion or evidence of cardiac failure
* moderate to severe renal insufficiency (creatinin clearance < 60 ml/min)
* psychogenic or habitual polydipsia
* hyponatraemia or predisposition for hyponatraemia
* diabetes insipidus
* syndrome of inadequate ADH production
* suspicion or evidence of liver failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-03-26 (Actual); Primary Completion 2013-02-01 (Actual); Study Completion 2015-02-01 (Actual)

PRIMARY OUTCOMES:
Blood samples for plasma concentration of Na+, K+, creatinin, osmolality (safety profile)at day 3. | At day 3 after first desmopressin intake.
Urine sample for urine concentration of Na+, K+, creatinin and osmolality | At day 3
Area Under Curve (AUC) frequency/volume chart during the first 14 days | Every day during the first 14 days.
The decrease of number of nocturnal micturition episodes. | At day 0
  Questionnaires at day 0 to evaluate the decrease of number of nocturnal micturition episodes.
The decrease of the number of nocturnal micturition episodes. | At day 30
  Questionnaires at day 30 to evaluate the number of nocturnal micturition episodes
Registration of number of side effects at day 3. | At day 3
Blood samples for plasma concentration of Na+, K+, creatinin, osmolality (safety profile)at day 7. | At day 7 after first desmopressin intake
Blood samples for plasma concentration of Na+, K+, creatinin, osmolality (safety profile)at day 30. | At day 30 after first desmopressin intake
Registration of number of side effects at day 7 | At day 7
Registration of number of side effects at day 30. | At day 30

CONTACTS AND LOCATIONS:
Overall Officials: Karel Everaert, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be